CLINICAL TRIAL: NCT02054169
Title: Pilot Study on the Feasibility of the Modified Confusion Assessment Method for the Emergency Department (mCAM-ED)
Brief Title: Feasibility of the Modified Confusion Assessment Method for the Emergency Department (mCAM-ED)
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Christian Nickel, MD, University Hospital, Basel, Switzerland
Other Study IDs: mCAM-ED
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- pre-test group: All patients aged 65 or older presenting to the ED during the pre-test period
- post-test period: All patients aged 65 or older presenting to the ED in the post-test period

SUMMARY:
Delirium is common in older emergency department (ED) patients and often remains unrecognized. Existing instruments to detect delirium are often time consuming and therefore not feasible in the busy ED setting In this study the investigators tested the feasibility of the newly developed modified confusion assessment method (mCAM-ED).

ELIGIBILITY:
Inclusion Criteria:

* patients aged 65 or older

Exclusion Criteria:

* patients treated in the resuscitation room
* patients transferred or discharged within 2 hours of arrival
* patients with insufficient proficiency in the German language
* patients with an inability to communicate (e.g. aphasic patients)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The samples consisted of consecutive ED patients.
Sampling Method: Probability Sample
Enrollment: 340 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
delirium | two hours after ED admission
  Delirium was assessed by research assistants using the mCAM-ED. Patients with a positive delirium diagnosis were presented to a senior emergency physician (PI) who served as the reference standard. The final delirium diagnosis was based on the DSM IV criteria

SECONDARY OUTCOMES:
adherence of ED staff to mCAM-ED algorithm | At patient discharge or transfer from ED (average 4 hours after presentation)
  Adherence was achieved when the mCAM-ED result was documented by the ED nurses.

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Nickel, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland